CLINICAL TRIAL: NCT01388452
Title: Presumptive and Definitive Virologic HIV Diagnosis in Hospitalized Malawian Infants
Brief Title: HIV Diagnosis in Hospitalized Malawian Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Fogarty International Center of the National Institute of Health (NIH); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 10-0441; R24TW007988 (NIH); 5P30AI050410 (NIH)
Record Dates: First submitted 2011-06-14; First posted 2011-07-06 (Estimated); Last update posted 2013-05-14 (Estimated); Status verified 2013-05

CONDITIONS: HIV Infections
Keywords: HIV; routine HIV testing; provider-initiated HIV testing and counseling; early infant diagnosis; Africa South of the Sahara
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Point of Care HIV RNA PCR (Experimental): Patients randomized to this arm will be followed prospectively from the time of clinical evaluation in the hospital until 12 months after returning for outpatient care at the KCH HIV clinic. The counselor will collect infant blood for point of care RNA PCR testing, number the sample, and transport it to the central laboratory for processing. Patients determined to be HIV-uninfected or HIV-exposed uninfected will not continue in the study beyond virologic test result disclosure, which will occur as an inpatient at KCH for this arm. If the patient does not return for outpatient care for three months after hospitalization then the patient's participation in the study will end.
  Interventions: Device: Point of care HIV RNA PCR
- Standard of Care (No Intervention): Patients randomized to this arm will be followed prospectively from the time of clinical evaluation in the hospital until 12 months after returning for outpatient care at the KCH HIV clinic. The counselor will collect infant blood for dried blood spot DNA PCR testing, number the sample, and transport it to the central laboratory for processing. If the patient is PD positive then the patient will be offered ART initiation prior to hospital discharge.
  Patients determined to be HIV-uninfected or HIV-exposed uninfected will not continue in the study beyond virologic test result disclosure, which will occur as an outpatient at KCH for this arm. If the patient does not return for outpatient care for three months after hospitalization then the patient's participation in the study will end.

INTERVENTIONS:
Device: Point of care HIV RNA PCR — The intervention is a HIV RNA PCR test for which UNC Project laboratory personnel will process samples in 48 hours so that patients can receive results prior to hospital discharge.
  Arms: Point of Care HIV RNA PCR

SUMMARY:
Purpose: The purpose of this research study is to learn about two HIV tests - a clinical "presumptive diagnosis" (PD) that a trained healthcare provider can quickly use to determine if a child is likely to be HIV-infected and in need of HIV medicines and an "expedited" gold standard RNA-PCR test (expedited PCR) that is done at the UNC Project lab located at the hospital and the result given within 48 hours. Both of these tests can obtain results quickly while the current test called dried blood spot DNA-PCR goes to a lab and the result may take up to one month. The performance of PD and expedited PCR will be compared to one another with respect to HIV-infected infants correctly initiating life-saving antiretroviral therapy.

Participants: Hospitalized children younger than 12 months of age who are HIV DNA-PCR eligible at Kamuzu Central Hospital (KCH), in Lilongwe, Malawi. Other participants will be patient caregivers and clinical officers who provide healthcare for children that could be HIV-infected. Clinical officers will be trained to conduct the presumptive diagnosis test.

Procedures (methods): Patients will be randomized to either standard of care (PD and dried blood spot DNA-PCR) or expedited PCR. A consultant pediatrician and a clinical officer will perform the PD. If the PD or expedited PCR test results are positive, hospital care could include HIV medicine.

DETAILED DESCRIPTION:
Background A majority of HIV-infected children die by two years of age without antiretroviral therapy (ART). Unfortunately, diagnosing HIV in this age group is complex as it requires virologic testing. This has served as a barrier to younger HIV-infected (HIV+) children accessing ART in resource-constrained generalized epidemic countries. Malawi, a high HIV-prevalence country in sub-Saharan Africa, implemented a national early infant diagnosis (EID) program utilizing virologic testing with dried blood spots (DBS) DNA PCR technology in 2007 to address this gap.

In coordination with the national EID program in 2008, we implemented a routine HIV testing strategy within the pediatric inpatient ward at Kamuzu Central Hospital (KCH) that incorporated DBS. While our initial program results have been encouraging, we have observed that only 50.2% of DBS recipients have returned for their test results after hospital discharge, draining resources and reducing the potential impact of definitive virologic testing and early diagnosis. DBS technology is a contributing factor to low patient follow-up as it requires burdensome transport and lengthy processing by highly trained laboratory personnel, requiring patients to return several weeks after testing for their results. Currently in Malawi, as is the case throughout sub-Saharan Africa, definitive virologic testing that provides test results prior to hospital discharge is not routinely available.

Two alternatives that could potentially strengthen EID and pediatric ART access are the routine use of presumptive diagnosis (PD), or a clinical HIV diagnostic algorithm in young children, as an adjunct to DBS and definitive inpatient virologic testing that provides results before hospital discharge ("expedited PCR") instead of PD and DBS. This research proposal primarily aims to validate PD testing as well as assess the impact of PD and expedited PCR upon patient outcomes within the established inpatient pediatric HIV testing system at KCH.

RESEARCH QUESTION TO BE ADDRESSED BY THIS PROPOSAL Is presumptive diagnosis, as an adjunct to dried blood spot DNA PCR, a valid approach for diagnosing HIV in hospitalized Malawian children younger than 12 months of age, and how does this strategy, compared to an expedited inpatient virologic diagnosis, affect patient outcomes?

RATIONALE FOR RESEARCH

Globally, an estimated 2.2 million children younger than 15 years of age were HIV-infected in 2007, with approximately 90% living in sub-Saharan Africa. Malawi, a sub-Saharan African country of 13.2 million people, reports an adult HIV prevalence of 11.9%. While 91,000 HIV+ children were estimated to be living in Malawi in 2007, less than 8% of all Malawian children have ever been HIV tested. Additionally, HIV+ children comprised just 8% of all national ART recipients, well below the 2014 goal of 15%. To address this gap, Malawi approved the routine offering of HIV testing, or provider initiated HIV testing and counseling (PITC), in line with global recommendations in 2007. While there is a high HIV prevalence in hospitalized Malawian children and current guidelines support routine inpatient HIV testing, no clear implementation strategy for hospitals has been offered.

Substantial percentages of HIV+ infants suffer from high mortality without early infant diagnosis (EID) and ART initiation, irrespective of CD4%, leading to the recommendation that all HIV+ children younger than 1 year of age should be universally initiated on ART. Despite the simplification of ART eligibility in this age group, diagnosing HIV remains complex. Maternal HIV antibodies can circulate in the blood stream of children until 12 months of age, confounding HIV antibody test results unable to discriminate between the mother's and child's antibodies. Accordingly, DNA PCR testing that detects HIV proviral DNA is the gold standard for HIV diagnosis in this age group. To date the PCR technology utilized in EID programs throughout sub-Saharan Africa, including Malawi, is DBS. Malawi piloted an EID program starting in 2007 and approved a policy of universal ART for all HIV+ children younger than 1 year of age in 2008. In Malawi, a uniform first line fixed-dose combination ART regimen of stavudine, lamivudine, and nevirapine is provided free of charge by the Malawian government for all eligible patients.The EID program has since expanded to 14 of 28 districts. Importantly, the national EID program identified the pediatric inpatient wards as a critical access point for routine DBS testing, but recently reported that few EID sites have established routine inpatient testing programs.

KCH is a referral hospital with a 215 bed pediatric ward located in the capital of Lilongwe with more than 10,000 pediatric admissions annually. In 2007, less than 10% of pediatric inpatients at KCH were estimated to have accessed voluntary HIV counseling and testing (VCT) services offered by lay counselors (Pediatric Department, KCH, unpublished data). In January 2008, we implemented a PITC program utilizing DBS testing in the KCH inpatient pediatric department in collaboration with the Baylor International Pediatric AIDS Initiative (BIPAI), KCH, and Lighthouse. The overall program objectives were to improve inpatient pediatric HIV diagnosis and care, establish EID as a routine inpatient service, and provide national guidance for inpatient pediatric PITC program expansion.

Over the first 12 months of implementation, the PITC program offered HIV testing to 45.2% of admissions, or 10,245 mothers and their hospitalized children, representing a four-fold increase in comparison to pre-PITC estimates1. 98.7% of mother-child pairs accepted testing, and we observed the HIV prevalence of hospitalized children to be 8.5%, nearly two-fold higher than the estimated community pediatric prevalence of 4.8% in Malawi. Furthermore, 73.9% of HIV+ hospitalized children had not yet accessed ART , despite over 70% of these patients clinically or immunologically eligible. The program also completed 476 DBS tests during the same time period, representing the highest volume EID site in Malawi, with 40.1% testing positive.

Unfortunately, only 239 DBS recipients, or 50.2% of children tested, enrolled into outpatient care at the Baylor College of Medicine-Abbott Fund Children's Clinical Centre of Excellence clinic at KCH. Of these, 48.3% were initiated on ART a median of 2.4 months after DBS collection. Low follow-up has been experienced at other EID sites throughout Malawi. One contributing factor is the several weeks of processing time required for DBS samples. In Malawi, DBS tests are transported to and from central laboratories to be processed in higher volumes by sophisticated equipment and highly specialized laboratory personnel. Therefore, counselors instruct caregivers to return in at least one month for their child's DBS test results. If caregivers return for their child's results, they are then commonly re-referred for HIV care at another site, often at an even later date, further delaying evaluation for ART eligibility. Currently, a similar system exists at KCH. Despite substantial investment into EID, the processing and transport delays inherent to DBS have lessened the impact of EID and have resulted in a continued barrier to pediatric ART access in this age group.

Two diagnostic alternatives that could reduce the delays complicating the current DBS systems are PD and point of care virologic testing. While PD is a less sensitive and specific diagnostic alternative to PCR, it requires limited resources and provides a strategy to immediately offer ART to hospitalized patients that fulfill PD criteria, avoiding the one-month wait time and resultant losses to follow-up. Malawi National guidelines recommend the use of PD to identify and initiate symptomatic HIV+ infants younger than 12 months of age on ART when PCR is unavailable. While the sensitivity and specificity of PD has been previously reported from Rwanda and Kenya, these studies are only partly applicable to Malawi due to the lower estimated malaria burdens in Rwandese children, and the mixture of inpatients and outpatients within the Kenyan study cohort. Both scenarios are likely to alter the reported sensitivities and specificities of PD as compared to Malawi, justifying the need to generate locally applicable data. To date, PD has not been widely practiced in Malawi, and data generated from this research could provide guidance to increase the usefulness of PD. The primary limitation to PD is that HIV-uninfected patients could be incorrectly started on ART. However, it is possible that such patients might still experience lower mortality and HIV transmission rates, with little adverse effects, as suggested by the recent outcomes of extended post-natal antiretroviral prophylaxis studies.

Point of care virologic testing, on the other hand, has the potential to revolutionize pediatric HIV care as HIV+ hospitalized infants could receive same day, accurate diagnostic results, allowing immediate evaluation for ART eligibility and initiation. While no point of care virologic test has yet been approved for routine use, the enhanced laboratory services available at University of North Carolina Project (UNC Project) can offer HIV RNA PCR test results in less than 48 hours. "Expedited" virologic testing is likely to provide definitive HIV test results to nearly all hospitalized HIV-exposed infants prior to discharge, therefore replicating the affect that point of care virologic testing will produce in the hospitalized setting. Understanding how expedited PCR testing affects inpatient ART uptake, outpatient follow-up, and longer term outcomes, compared to the current standard of care, will be critical for further system development and strengthening in anticipation of future point of care test availability.

This research proposal seeks to utilize the current inpatient pediatric PITC system established at KCH to validate PD within the hospital setting, as well as investigate patient outcomes utilizing current EID standard of care (PD and DBS) compared to expedited PCR.

ELIGIBILITY:
Inclusion Criteria:

* Male and female children
* Less than 12 months of age
* Inpatient at KCH
* HIV DNA-PCR test eligible
* No prior definitive PCR test result

Exclusion Criteria:

* Caregiver does not want to be contacted by study team
* Mother initiated on ART prior to pregnancy

Max Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Actual)
Dates: Start 2011-06; Primary Completion 2011-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
ART initiation of HIV-infected infants | Participants will be followed for an expected average of 2 months, or until their HIV-status is confirmed
  The primary outcome will be the proportion of HIV+ children initiated on ART in the hospital. We will need a sample size of 400 infants assuming the standard of care will initiate 60% and the experimental group will initiate 85% of HIV-infected infants on ART prior to hospital discharge, respectively. These assumptions also take into consideration a predicted inpatient HIV-prevalence in HIV-exposed infants of 25% and a 5% absconding rate, using a confidence interval of 10% and confidence level of p < 0.05.

CONTACTS AND LOCATIONS:
Overall Officials: Eric D McCollum, MD, Principal Investigator — UNC Project; Mina Hosseinipour, MD, MPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Kamuzu Central Hospital, Lilongwe, Malawi

REFERENCES:
- [Background] 1. Joint United Nations Programme on HIV/AIDS (2008) 2008 Report on the Global AIDS Epidemic. Available: http://data.unaids.org/pub/GlobalReport/2008/JC1511_GR08_ExecutiveSummary_en.pdfAccessed 7 September 2009.
- [Background] 2. The United Nations Children's Fund (2008) Children and AIDS: Third Stocktaking Report, 2008. Available: http://www.unicef.org/publications/index_46585.html. Accessed 7 September 2009.
- [Background] 3. Ministry of Health Malawi: HIV Unit (2008) Annual Report HIV Unit 2008.
- [Background] 4. World Health Organization (2007) Guidance on provider-initiated HIV testing and counseling in health facilities. Available: http://whqlibdoc.who.int/publications/2007/9789241595568_eng.pdf. Accessed 26 August 2009.
- [Background] Rogerson SR, Gladstone M, Callaghan M, Erhart L, Rogerson SJ, Borgstein E, Broadhead RL. HIV infection among paediatric in-patients in Blantyre, Malawi. Trans R Soc Trop Med Hyg. 2004 Sep;98(9):544-52. doi: 10.1016/j.trstmh.2003.12.011. PMID 15251404
- [Background] 6. Ministry of Health Malawi: HIV Unit (2008) Guidelines for Paediatric HIV Testing and Counseling.
- [Background] Violari A, Cotton MF, Gibb DM, Babiker AG, Steyn J, Madhi SA, Jean-Philippe P, McIntyre JA; CHER Study Team. Early antiretroviral therapy and mortality among HIV-infected infants. N Engl J Med. 2008 Nov 20;359(21):2233-44. doi: 10.1056/NEJMoa0800971. PMID 19020325
- [Background] Diaz C, Hanson C, Cooper ER, Read JS, Watson J, Mendez HA, Pitt J, Rich K, Smeriglio V, Lew JF. Disease progression in a cohort of infants with vertically acquired HIV infection observed from birth: the Women and Infants Transmission Study (WITS). J Acquir Immune Defic Syndr Hum Retrovirol. 1998 Jul 1;18(3):221-8. doi: 10.1097/00042560-199807010-00004. PMID 9665498
- [Background] Tovo PA, de Martino M, Gabiano C, Cappello N, D'Elia R, Loy A, Plebani A, Zuccotti GV, Dallacasa P, Ferraris G, et al. Prognostic factors and survival in children with perinatal HIV-1 infection. The Italian Register for HIV Infections in Children. Lancet. 1992 May 23;339(8804):1249-53. doi: 10.1016/0140-6736(92)91592-v. PMID 1349667
- [Background] Newell ML, Coovadia H, Cortina-Borja M, Rollins N, Gaillard P, Dabis F; Ghent International AIDS Society (IAS) Working Group on HIV Infection in Women and Children. Mortality of infected and uninfected infants born to HIV-infected mothers in Africa: a pooled analysis. Lancet. 2004 Oct 2-8;364(9441):1236-43. doi: 10.1016/S0140-6736(04)17140-7. PMID 15464184
- [Background] Chilongozi D, Wang L, Brown L, Taha T, Valentine M, Emel L, Sinkala M, Kafulafula G, Noor RA, Read JS, Brown ER, Goldenberg RL, Hoffman I; HIVNET 024 Study Team. Morbidity and mortality among a cohort of human immunodeficiency virus type 1-infected and uninfected pregnant women and their infants from Malawi, Zambia, and Tanzania. Pediatr Infect Dis J. 2008 Sep;27(9):808-14. doi: 10.1097/INF.0b013e31817109a4. PMID 18679152
- [Background] Dunn D; HIV Paediatric Prognostic Markers Collaborative Study Group. Short-term risk of disease progression in HIV-1-infected children receiving no antiretroviral therapy or zidovudine monotherapy: a meta-analysis. Lancet. 2003 Nov 15;362(9396):1605-11. doi: 10.1016/s0140-6736(03)14793-9. PMID 14630440
- [Background] 13. World Health Organization (2006) Report of the WHO Technical Reference Group, Paediatric HIV/ ART Care Guideline Group Meeting.
- [Background] 14. World Health Organization (2006) Antiretroviral therapy of HIV infection in infants and children in resource-limited settings: towards universal access. Available: http://www.who.int/ hiv/pub/guidelines/pmtctguidelines3.pdf. Accessed 17 November 2009.
- [Background] Sherman GG, Cooper PA, Coovadia AH, Puren AJ, Jones SA, Mokhachane M, Bolton KD. Polymerase chain reaction for diagnosis of human immunodeficiency virus infection in infancy in low resource settings. Pediatr Infect Dis J. 2005 Nov;24(11):993-7. doi: 10.1097/01.inf.0000187036.73539.8d. PMID 16282936
- [Background] 16. United Nations Children's Fund (2008) Children and AIDS. Third Stocktaking Report, 2008. Available at: http:// www.unicef.org/publications. Accessed 17 November, 2009.
- [Background] 17. Ministry of Health Malawi and National AIDS Commission (2008) Treatment of AIDS: Guidelines for the Use of Antiretroviral Therapy in Malawi, Third Edition.
- [Background] 18. Ministry of Health Malawi and National AIDS Commission (2009) Early Infant Diagnosis Report, 24 August.
- [Background] 19. Kabue MM, Braun M, Aetker L, Chirwa M, Mofolo I, et al. (2009) ART initiation and increased survival of infants traced from PMTCT to pediatric HIV care: highlighting the need for program coordination in Lilongwe, Malawi. 5th Conference on HIV Pathogenesis, Treatment and Prevention. Cape Town, South Africa. Abstract WEPDD103.
- [Background] Peltier CA, Omes C, Ndimubanzi PC, Ndayisaba GF, Stulac S, Arendt V, Courteille O, Muganga N, Kayumba K, Van den Ende J. Validation of 2006 WHO prediction scores for true HIV infection in children less than 18 months with a positive serological HIV test. PLoS One. 2009;4(4):e5312. doi: 10.1371/journal.pone.0005312. Epub 2009 Apr 24. PMID 19390690
- [Background] Inwani I, Mbori-Ngacha D, Nduati R, Obimbo E, Wamalwa D, John-Stewart G, Farquhar C. Performance of clinical algorithms for HIV-1 diagnosis and antiretroviral initiation among HIV-1-exposed children aged less than 18 months in Kenya. J Acquir Immune Defic Syndr. 2009 Apr 15;50(5):492-8. doi: 10.1097/QAI.0b013e318198a8a4. PMID 19225401
- [Background] Kilewo C, Karlsson K, Massawe A, Lyamuya E, Swai A, Mhalu F, Biberfeld G; Mitra Study Team. Prevention of mother-to-child transmission of HIV-1 through breast-feeding by treating infants prophylactically with lamivudine in Dar es Salaam, Tanzania: the Mitra Study. J Acquir Immune Defic Syndr. 2008 Jul 1;48(3):315-23. doi: 10.1097/QAI.0b013e31816e395c. PMID 18344879
- [Background] Kumwenda NI, Hoover DR, Mofenson LM, Thigpen MC, Kafulafula G, Li Q, Mipando L, Nkanaunena K, Mebrahtu T, Bulterys M, Fowler MG, Taha TE. Extended antiretroviral prophylaxis to reduce breast-milk HIV-1 transmission. N Engl J Med. 2008 Jul 10;359(2):119-29. doi: 10.1056/NEJMoa0801941. Epub 2008 Jun 4. PMID 18525035
- [Background] Six Week Extended-Dose Nevirapine (SWEN) Study Team; Bedri A, Gudetta B, Isehak A, Kumbi S, Lulseged S, Mengistu Y, Bhore AV, Bhosale R, Varadhrajan V, Gupte N, Sastry J, Suryavanshi N, Tripathy S, Mmiro F, Mubiru M, Onyango C, Taylor A, Musoke P, Nakabiito C, Abashawl A, Adamu R, Antelman G, Bollinger RC, Bright P, Chaudhary MA, Coberly J, Guay L, Fowler MG, Gupta A, Hassen E, Jackson JB, Moulton LH, Nayak U, Omer SB, Propper L, Ram M, Rexroad V, Ruff AJ, Shankar A, Zwerski S. Extended-dose nevirapine to 6 weeks of age for infants to prevent HIV transmission via breastfeeding in Ethiopia, India, and Uganda: an analysis of three randomised controlled trials. Lancet. 2008 Jul 26;372(9635):300-13. doi: 10.1016/S0140-6736(08)61114-9. PMID 18657709
- [Background] 25. Chasela C, Hudgens M , Jamieson D , Kayira D , Hosseinipour M, et al. (2009) Both maternal HAART and daily infant nevirapine (NVP) are effective in reducing HIV-1 transmission during breastfeeding in a randomized trial in Malawi: 28 week results of the Breastfeeding, Antiretroviral and Nutrition (BAN) Study. 5th Conference on HIV Pathogenesis, Treatment and Prevention. Cape Town, South Africa. Abstract WELBC103.
- [Background] 26. World Health Organization (2008) World Malaria Report. Available: http://apps.who.int/malaria/wmr2008/malaria2008.pdf. Accessed 19 November 2009.